CLINICAL TRIAL: NCT00973570
Title: Evaluation of a Smoking Cessation Program Among ADOlescents in Vocational Training Centers
Brief Title: Smoking Cessation Program Among Adolescents in Vocational Training Centers
Acronym: TABADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: University of Nancy (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C07-43
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2009-09

CONDITIONS: Tobacco Use
Keywords: tobacco cessation; evaluation; epidémiology; adolescent; apprentices
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Intervention" group (Experimental): The "intervention" group benefits from the TABADO program
  Interventions: Behavioral: TABADO program
- "Control" group (No Intervention): The "control" group not benefit from any specific intervention other than the treatment and education usually available

INTERVENTIONS:
Behavioral: TABADO program — The intervention takes place in 3 stages: (i) a general information session on tobacco consumption is delivered to all teenagers, both smokers and nonsmokers. (ii) For smokers wishing to join the program, this session is followed by individualized consultations with a team of tobacco addiction physicians. (iii) The volunteers then benefit from a small group approach, consisting of discussion sessions to share experiences, strengthen motivation, and prevent relapse. There will be 4 sessions in total, comprising individual counseling and work in groups spread over 3 months (taking into account the availability of the trainees because of their alternate-week training schedule).
  Arms: "Intervention" group

SUMMARY:
Background: Most of the efforts to fight against young people's tobacco addiction have focused on smoking prevention and little on smoking cessation. A smoking cessation program, associating pharmacologic and cognitive-behavioural strategy, on a particularly vulnerable population (vocational trainees), was developed by a team of tobacco addiction specialist physicians. We developed a study to evaluate the efficacy of the program. Its main objective is to compare the efficacy of a smoking cessation program offered to all smokers in a population aged 15 to 20 years in Vocational Training Centers (VTC) with that in a control population. The objective of this paper is to present the TABADO study protocol and the results of the pilot study.

Methods: The study is quasi-experimental, prospective, evaluative and comparative and takes place during the 2 years of vocational training. The final population will be composed of 2000 trainees entering a VTC (in Lorraine, France): The intervention group (1000 trainees) benefited from the TABADO program while no specific intervention took place in the "control" group (1000 trainees) other than the treatment and education services usually available. Our primary outcome will be the tobacco abstinence rate at 12 months.

The pilot study is a descriptive monocentric cross-sectional study conducted among the whole group of students, completed by a longitudinal prospective study of smoker volunteers.

ELIGIBILITY:
Inclusion criteria:

* All students, males and females, registered in the VTC for at least a 2-year training period
* Aged from 15 to 20 years

Exclusion criteria:

* Subjects with current serious psychiatric disorders or who may be susceptible to decompensation upon quitting smoking (major depression)
* Smokers who are involved in an ongoing attempt to quit, with medical monitoring.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the rate of smoking abstinence after 12 months, measured on the basis of the statements of the whole sample, not only among volunteers. | 12 months

SECONDARY OUTCOMES:
Overall prevalence of tobacco use in the institutions concerned at 12 months. | 12 months
Students' motivation to quit smoking (motivational score) and frequency of attempts to quit within the 12 months after the intervention | 12 months
Rate of withdrawal from the program among the volunteers after 12 months. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: François ALLA, MD/ PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- CHU Nancy, Nancy, Lorraine, France

REFERENCES:
- [Background] Minary L, Martini H, Wirth N, Thouvenot F, Acouetey DS, Martinet Y, Bohadana A, Zmirou-Navier D, Alla F. TABADO: "evaluation of a smoking cessation program among adolescents in vocational training centers": study protocol. BMC Public Health. 2009 Nov 13;9:411. doi: 10.1186/1471-2458-9-411. PMID 19912627